CLINICAL TRIAL: NCT02959294
Title: Use of Adipose-Derived Cellular Stromal Vascular Fraction (AD-cSVF) Parenterally in Post-Concussion Injuries and Traumatic Brain Injuries (TBI)
Brief Title: Use of Adipose-Derived Stem/Stromal Cells in Concussion and Traumatic Brain Injuries
Acronym: C-TBI
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: COVID restrictions prevent patient enrollment or treatment. Clinical Trial facility is being closed due to viral limitations and loss of staff to perform]]
Sponsor: Robert W. Alexander, MD, FICS (Industry)
Responsible Party: Sponsor-Investigator, Robert W. Alexander, MD, FICS, Principal Investigator, Healeon Medical Inc
Organization: Healeon Medical Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGV GARM 5
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Encephalopathies, Chronic; Concussion, Mild; Concussion, Intermediate; Concussion, Severe; Concussion, Brain
Keywords: TBI; mTBI; Concussion, Brain; Loss Consciousness, Traumatic; Headaches
MeSH Terms: conditions — Brain Injuries, Traumatic; Bronchiolitis Obliterans Syndrome; Brain Concussion; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Microcannula Harvest Adipose (Experimental): Acquisition Adipose-Derived Tissue Stromal Vascular Fraction (AD-tSVF) via close syringe microcannula harvest from subdermal fat deposits
  Interventions: Procedure: Microcannula Harvest Adipose
- Centricyte 1000 (Experimental): Autologous AD-tSVF via enzymatic isolation/concentration via Centricyte 1000 Closed System to create AD-cSVF
  Interventions: Device: Centricyte 1000
- Sterile Normal Saline (Experimental): Re-suspension of AD-cSVF pellet in Normal Saline deployment via IV
  Interventions: Procedure: Sterile Normal Saline IV deployment AD-cSVF

INTERVENTIONS:
Procedure: Microcannula Harvest Adipose — Use of Closed Syringe Microcannula Harvest Autologous Adipose-Derived Stem/Stromal Cells
  Arms: Microcannula Harvest Adipose
Device: Centricyte 1000 — Use of Centricyte 1000 Closed System Digestion Autologous AD-tSVF to create AD-cSVF
  Arms: Centricyte 1000
Procedure: Sterile Normal Saline IV deployment AD-cSVF — Sterile Normal Saline Suspension AD-cSVF in 500 cc IV use
  Arms: Sterile Normal Saline

SUMMARY:
Concussion is the most common type of brain injury throughout life. Study is seeking improvement of long-term residua following adolescent and adult post-traumatic injuries often associated with contact sports and accidental causes. Typically defined as reversible head injury with temporary loss of brain function. Symptoms range from physical, cognitive, pain (headache) and emotional signs consistent with TBI and Post-Traumatic Stress Syndrome. Use of AD-cSVF parenteral delivery to encourage repair of damage and decreased function following concussion, particularly in contact, repetitive sports injuries. Range of damage is measured in Grade I-III according to graduated severity. Unfortunately, less information is available about repetitive concussions and the long-term health issues.

DETAILED DESCRIPTION:
Concussion Syndrome (CS) and TBI are common injuries producing temporary and long-term damage to impact brain function. Symptoms are sometimes transient, sometimes long-term depending on severity and/or repetitive damage. Signs varying from recurrent headaches, mental fog, emotional changes to physical signs of loss of consciousness, amnesia to behavioral change (irritability, loss of concentration ability, etc.), cognitive impairment (slow reaction times, memory loss), and recurring sleep disturbances.

Common causes include sports injuries, automobile accidents, falls, blunt trauma to head, and explosive/blast injuries from production of acceleration injuries

Treatment often involves monitoring, physical rest, limiting cognitive activities (such as computing, video games, texting, and studying). Most often a single episode usually resolve or improve (particularly in recurring headaches) within 3-4 weeks. It is estimated that >6/1000 occurrence rate apply. Repetitive injuries seem to make the person more susceptible to additional damage, particularly with injury precedes resolution of an earlier damage. There appears also to make persons to require a lesser impact to produce the same degree of severity. It is becoming more recognized that repeated concussions increase the risks in later life for dementia, Parkinson's and severe depressions.

Most serious signs to evaluate are loss of consciousness, seizures, worsening headache, diplopia/pupil changes, loss of recognition, vomiting, focal neurological problems, and change of personality.

There is no consensus definition of concussion or TBI. Most concussions are considered in the mild TBI (mTBI) group, and are rarely demonstrate structural brain damage when in the acute to subacute state. Late brain MRI changes are difficult to clearly point to or identify the specific areas of presumed damage.

This study is intended to examine safety and efficacy of parenteral introduction of AD-cSVF in cases of CS and TBI, and categorically examine the outcomes according to the elapsed time from original concussive event. No delineation of those having recurrent damage and injuries are made within this study.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of mTBI or TBI with Correlated MRI or CT
* At least 1 month post mTBI and TBI
* Able and Willing to participate in CT or MRI pre-study and at 3 year, 5 year interval
* Able to provide informed consent to undergo the study
* Depression, Cognitive Disability, Attention Disorders, Headaches or other persistent changes which followed a traumatic brain event (TBI)
* Impaired social or occupational functioning following mTBI or TBI
* History of repetitive events for mTBI and TBI

Exclusion Criteria:

* Documented history of neuro-degenerative illness, seizures, mental illness, or severe medical conditions preceding mTBI or TBI
* Malignances, Bleeding Disorders, Pregnancy or Lactation
* Tumors of Central Nervous System (CNS)
* Lack of adequate donor tissue volume as determined by the primary investigator at their discretion
* Any pre-existing medical condition which, in view of the primary investigator and patient's primary care physician, would prevent participation in study

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | Outcome measures at baseline at 6 month
  Activities of Daily Living (ADL)
Cognitive Change in clinical symptoms associated with concussion-TBI | Outcome measures at baseline and reviewed 1 year interval for average time 5 years
  Montreal Cognitive Assessment Scale (MCAS)

SECONDARY OUTCOMES:
Beck's Depression Inventory (BDI) | Annual for 5 years
  Multiple choice self reporting measure of depression
Adult Attention Deficit Assessment | Annual for 5 years
  Conner's Adult Attention Deficit Disorder Rate Scale (CAADDR)
MRI Brain With & MRI Brain With & Without Contrast | 0, 3 years, 5 years
  MRI Brain to evaluate progressive changes comparing pre-treatment (0), 3 year and 5 year status

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Alexander, MD, Principal Investigator — GARM International and GARM USA; Glenn C Terry, MD, Principal Investigator — GARM
Locations (1):
- Regenevita LLC, Stevensville, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Annual Summary of Case to All Collaborators

REFERENCES:
- [Background] Maas AI, Stocchetti N, Bullock R. Moderate and severe traumatic brain injury in adults. Lancet Neurol. 2008 Aug;7(8):728-41. doi: 10.1016/S1474-4422(08)70164-9. PMID 18635021
- [Background] Parikh S, Koch M, Narayan RK. Traumatic brain injury. Int Anesthesiol Clin. 2007 Summer;45(3):119-35. doi: 10.1097/AIA.0b013e318078cfe7. No abstract available. PMID 17622833
- [Background] Saatman KE, Duhaime AC, Bullock R, Maas AI, Valadka A, Manley GT; Workshop Scientific Team and Advisory Panel Members. Classification of traumatic brain injury for targeted therapies. J Neurotrauma. 2008 Jul;25(7):719-38. doi: 10.1089/neu.2008.0586. PMID 18627252
- [Background] Kumar R, Husain M, Gupta RK, Hasan KM, Haris M, Agarwal AK, Pandey CM, Narayana PA. Serial changes in the white matter diffusion tensor imaging metrics in moderate traumatic brain injury and correlation with neuro-cognitive function. J Neurotrauma. 2009 Apr;26(4):481-95. doi: 10.1089/neu.2008.0461. PMID 19196176
- [Background] Pellman EJ, Viano DC; National Football League's Committee on Mild Traumatic Brain Injury. Concussion in professional football: summary of the research conducted by the National Football League's Committee on Mild Traumatic Brain Injury. Neurosurg Focus. 2006 Oct 15;21(4):E12. doi: 10.3171/foc.2006.21.4.13. PMID 17112190
- [Background] Heegaard W, Biros M. Traumatic brain injury. Emerg Med Clin North Am. 2007 Aug;25(3):655-78, viii. doi: 10.1016/j.emc.2007.07.001. PMID 17826211
- [Background] Pearce JM. Observations on concussion. A review. Eur Neurol. 2008;59(3-4):113-9. doi: 10.1159/000111872. Epub 2007 Nov 30. PMID 18057896
- [Background] Concussion (mild traumatic brain injury) and the team physician: a consensus statement. Med Sci Sports Exerc. 2005 Nov;37(11):2012-6. doi: 10.1249/01.mss.0000186726.18341.70. No abstract available. PMID 16286874
- [Background] Hall RC, Hall RC, Chapman MJ. Definition, diagnosis, and forensic implications of postconcussional syndrome. Psychosomatics. 2005 May-Jun;46(3):195-202. doi: 10.1176/appi.psy.46.3.195. PMID 15883140
- [Background] Maroon JC, Lovell MR, Norwig J, Podell K, Powell JW, Hartl R. Cerebral concussion in athletes: evaluation and neuropsychological testing. Neurosurgery. 2000 Sep;47(3):659-69; discussion 669-72. doi: 10.1097/00006123-200009000-00027. PMID 10981754
- [Background] Randolph C. Baseline neuropsychological testing in managing sport-related concussion: does it modify risk? Curr Sports Med Rep. 2011 Jan-Feb;10(1):21-6. doi: 10.1249/JSR.0b013e318207831d. PMID 21228656
- [Background] Binder LM. Persisting symptoms after mild head injury: a review of the postconcussive syndrome. J Clin Exp Neuropsychol. 1986 Aug;8(4):323-46. doi: 10.1080/01688638608401325. PMID 3091631
- [Background] Thornton KE, Carmody DP. Efficacy of traumatic brain injury rehabilitation: interventions of QEEG-guided biofeedback, computers, strategies, and medications. Appl Psychophysiol Biofeedback. 2008 Jun;33(2):101-24. doi: 10.1007/s10484-008-9056-z. Epub 2008 Jun 13. PMID 18551365
- [Background] Alexander MP. Mild traumatic brain injury: pathophysiology, natural history, and clinical management. Neurology. 1995 Jul;45(7):1253-60. doi: 10.1212/wnl.45.7.1253. No abstract available. PMID 7617178
- [Background] De Beaumont L, Theoret H, Mongeon D, Messier J, Leclerc S, Tremblay S, Ellemberg D, Lassonde M. Brain function decline in healthy retired athletes who sustained their last sports concussion in early adulthood. Brain. 2009 Mar;132(Pt 3):695-708. doi: 10.1093/brain/awn347. Epub 2009 Jan 28. PMID 19176544
- [Background] Cantu RC. Chronic traumatic encephalopathy in the National Football League. Neurosurgery. 2007 Aug;61(2):223-5. doi: 10.1227/01.NEU.0000255514.73967.90. No abstract available. PMID 17762733
- [Background] Jordan BD. Chronic traumatic brain injury associated with boxing. Semin Neurol. 2000;20(2):179-85. doi: 10.1055/s-2000-9826. PMID 10946737
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Cantu RC. Second-impact syndrome. Clin Sports Med. 1998 Jan;17(1):37-44. doi: 10.1016/s0278-5919(05)70059-4. PMID 9475969
- [Background] Borg J, Holm L, Peloso PM, Cassidy JD, Carroll LJ, von Holst H, Paniak C, Yates D; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Non-surgical intervention and cost for mild traumatic brain injury: results of the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):76-83. doi: 10.1080/16501960410023840. PMID 15083872